CLINICAL TRIAL: NCT03368170
Title: A Randomized, Placebo-controlled, Phase IIa Study Evaluating the Efficacy and Tolerability of IRL790 in Parkinson's Disease Dyskinesia
Brief Title: Efficacy and Tolerability of IRL790 in Parkinson's Disease Dyskinesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Integrative Research Laboratories AB (Industry)
Collaborators: The Clinical Trial Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRL790C003
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Results first posted 2020-03-24 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Parkinson Disease
Keywords: Levodopa induced dyskinesia
MeSH Terms: conditions — Parkinson Disease | interventions — mesdopetam

STUDY DESIGN:
Intervention Model Description: Double blind, placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesdopetam (IRL790) (Experimental): Capsule 2.5 mg, oral administration
  Interventions: Drug: Mesdopetam (IRL790)
- Placebo (Placebo Comparator): Identical capsule, oral administration
  Interventions: Drug: Mesdopetam (IRL790)

INTERVENTIONS:
Drug: Mesdopetam (IRL790) — Mesdopetam (IRL790) capsule
  Other Names: IRL790

SUMMARY:
Mesdopetam (IRL790) is an experimental small molecule compound with psychomotor stabilizing properties. The primary target is the dopamine D3 receptor, a target implicated in the generation of levodopa-induced dyskinesia, a side-effect frequently occurring with long-term levodopa treatment in patients with Parkinson's disease. In experimental animals mesdopetam potently reduced levodopa-induced involuntary movement without impairing the antiparkinsonian effect of levodopa.

The primary purpose of the trial is to investigate whether mesdopetam given as adjunctive treatment can reduce levodopa induced dyskinesia in patients with Parkinson's disease. The trial will also help to establish the most optimal dosing of the compound.

DETAILED DESCRIPTION:
METHODOLOGY:

This is a multicentre study where 74 patients with Parkinson's disease exhibiting levodopa induced dyskinesia will be randomised to receive study drug or placebo. Thirty seven patients will be randomised to mesdopetam and 37 patients to placebo (1:1 randomisation).

Patients will be screened for eligibility according to inclusion/exclusion criteria within four weeks of initiation of study treatment (Screening visit).

An outpatient study with the patients taking the study drug for four weeks at home. Mesdopetam will be taken twice daily (b.i.d.) as adjunctive treatment to the patients' regular and stable antiparkinsonian medication.

The first two weeks of treatment will allow for per patient titration of study medication to the highest tolerated predefined dose, after which patients will continue on this highest tolerated dose for an additional two weeks.

Changes in disease state and dyskinesia will be measured using the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) and Unified Dyskinesia Rating Scale (UDysRS); furthermore, patients will administer two 24-hour diaries on run-in and on the fourth week of dosing to assess daily movements.

Pharmacokinetic (PK) samples will be collected for the determination of concentrations of mesdopetam and its metabolites IRL902 and IRL872 in plasma. They will be collected before and after IMP administration at two visits.

A Follow-up Visit will be performed for all patients five to eight days after last administration of IMP.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥18 and ≤79 years of age.
2. Signed a current Ethics Committee approved informed consent form.
3. Parkinson's disease, per UK Parkinson's Disease Society (UKPDS) Brain Bank Clinical Diagnostic Criteria.
4. Waking day dyskinesia of ≥25% determined as a score of ≥2 as per Question 4.1 of the MDS-UPDRS.
5. On a stable regimen of antiparkinson medications for at least 30 days prior to screening, including a levodopa preparation administered not less than three times daily and willing to continue the same doses and regimens during study participation. Rescue medication such as Madopar dispersable and Apomorphine injections are allowed.
6. Taking a maximum of eight regular levodopa intakes per day, excluding bedtime and night time levodopa.
7. Any other current and allowed prescription/non-prescription medications and/or nutritional supplements taken regularly must have been at a stable dose and regimen for at least 30 days prior to screening and the patient must be willing to continue the same doses and regimens during study participation (this criterion does not apply to medications that are being taken pre-study only on an as-needed basis).
8. Patient must be willing and able to avoid direct exposure to sunlight from day 1 to day 28.
9. Able to complete at least one valid 24-hour patient diary at Visit 1.

Exclusion Criteria:

1. History of neurosurgical intervention related to Parkinson's disease (e.g. deep brain stimulation).
2. Treatment with pump delivered antiparkinsonian therapy (i.e. subcutaneous apomorphine or levodopa/carbidopa intestinal infusion).
3. History of seizures within two years prior to screening.
4. History of stroke or transient ischemic attack (TIA) within two years prior to screening.
5. History of cancer within five years prior to screening, with the following exceptions: adequately treated non-melanomatous skin cancers, localised bladder cancer, non-metastatic prostate cancer or in situ cervical cancer.
6. Presence of cognitive impairment, as evidenced by a Mini-Mental Status Examination (MMSE) score of less than 24 during screening.
7. A Hoehn and Yahr score of five when "off" as per Question 3.18 of the MDS-UPDRS, assessed during screening.
8. Any history of a significant heart condition or cardiac arrhythmias within the past 5 years, any repolarisation deficits or any other clinically significant abnormal ECG as judged by the Investigator
9. Severe or ongoing unstable medical condition including a history of poorly controlled diabetes; obesity associated with metabolic syndrome; uncontrolled hypertension; cerebrovascular disease, or any form of clinically significant cardiac disease; clinically significant symptomatic orthostatic hypotension; clinically significant hepatic disease, renal failure or abnormal renal function.
10. Any history of a neurological other than Parkinson's disease or a psychiatric disorder, including history of DSM IV diagnosed major depression or psychosis. Patients with illusions or hallucinations with no loss of insight will be eligible. Patients with mild depression who are well controlled on a stable dose of an antidepressant medication for at least 4 weeks before screening will be eligible.
11. Enrolment in any other clinical study involving medication, medical devices or surgical procedures, current or within three months prior to screening visit, or previous participation in the present study. Patients enrolled in non-interventional clinical trials will be eligible.
12. Drug and/or alcohol abuse.
13. History of severe drug allergy or hypersensitivity.
14. If female, is pregnant or lactating, or has a positive pregnancy test result pre-dose.
15. Patients unwilling to use two forms of contraception 90 days for men and 30 days for women after last IMP dose
16. Any planned major surgery within the duration of the study.
17. Any other condition or symptoms preventing the patient from entering the study, according to the Investigator's judgement.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Carroll, MD, Principal Investigator — Plymouth University Peninsula Schools of Medicine and Dentistry
Locations (20):
- Sweden (4):
  - Sahlgrenska University hospital, Gothenburg
  - University hospital, Linköping
  - University hospital, Lund
  - Karolinska University hospital, Stockholm
- United Kingdom (16):
  - Bristol Brain Centre, Southmead Hospital, Bristol
  - Fairfield General Hospital (Pennine Acute NHS Trust), Bury
  - Ninewells Hospital, Dundee
  - Lincoln County Hospital, Lincoln
  - Charing Cross Hospital, Imperial College Healthcare NHS Trust, London
  - The National Hospital of Neurology and Neurosurgery (UCL), London
  - Luton and Dunstable University Hospital NHS Foundation Trust, Luton
  - North Tyneside General Hospital, North Shields
  - Qeens' Medical Centre, Nottingham
  - John Radcliffe Hospital, Oxford
  - Peterborough City Hospital, Peterborough
  - Plymouth Hospitals NHS Trust - Derriford Hospital, Plymouth
  - Queens's Hospital, Romford
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Torbay hospital, Torquay
  - Royal Cornwall Hospital, Truro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McFarthing K, Prakash N, Simuni T. CLINICAL TRIAL HIGHLIGHTS - DYSKINESIA. J Parkinsons Dis. 2019;9(3):449-465. doi: 10.3233/JPD-199002. No abstract available. PMID 31356217

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted as an outpatient trial and patients were identified from 20 sites across two countries. The first patient was enrolled 13 April 2018 and the last past completed 12 June 2019.
Pre-assignment Details: Patients completed two 24-hour diaries during run-in of which one had to be valid prior randomization.
Groups:
- Mesdopetam: Mesdopetam capsule, 2.5 mg oral administration. Dose given twice daily (5 mg, 7.5 mg or 10 mg b.i.d.) The first two weeks of treatment allowed for per patient titration of study medication to the highest tolerated predefined dose, after which patients continued on this highest per patient tolerated dose for an additional two weeks.
- Placebo: Matching placebo capsule, oral administration. Dose given twice daily.
  The first two weeks of treatment allowed for per patient titration of study medication to the highest tolerated number of placebo capsules (1 capsule x 4), after which patients continued on this highest tolerated dose for an additional two weeks.
Period: Overall Study
Arm/Group | Mesdopetam | Placebo
Started | 39 | 36
Completed | 37 | 35
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Mesdopetam: Mesdopetam (IRL790): 2.5 mg white hard HPMC capsule, oral administration
- Placebo: Placebo: Matching placebo capsule, white hard HPMC capsule, oral administration
- Total: Total of all reporting groups
Arm/Group | Mesdopetam | Placebo | Total
Number analyzed (Participants) | 39 | 36 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (8.9) | 67.7 (7.7) | 66.6 (8.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 13 | 33
  Male | 19 | 23 | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 39 | 35 | 74
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 38 | 35 | 73
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.6 (7.2) | 25.3 (4.2) | 26 (5.92)
Height [Mean (Standard Deviation); unit: centimeters] | 166.7 (10.3) | 169 (9.4) | 168 (9.87)
Years with Parkinson's disease [Mean (Standard Deviation); unit: years] | 10.7 (5.9) | 10.7 (4.3) | 10.7 (5.15)

OUTCOME MEASURES:

1. Primary Outcome: Unified Dyskinesia Rating Scale (UDysRS)
Description: The change from baseline to day 28 of treatment (Visit 4) in the sum of the items comprising the Unified Dyskinesia Rating Scale (UDysRS). The Unified Dyskinesia Rating Scale (UDysRS) is administered to assess dyskinesia. The scoring range is 0-104, where higher score means more dyskinesia.
Time Frame: Baseline and 4 weeks
Population: Full analysis set (all randomized and treated patients who received one or more doses and who provided post baseline data whether or not they fully complied with the requirements of the protocol).
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Mesdopetam: Mesdopetam: 2.5 mg white hard HPMC capsule, oral administration
Arm/Group | Mesdopetam | Placebo
Number analyzed (Participants) | 36 | 34
score on a scale | -4.2 [-7.3 to -1.0] | -7.0 [-10.3 to -3.8]

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV, Question 4.1 and 4.2
Description: Change in MDS-UPDRS sum score of questions 4.1 (Time spent with dyskinesias) and 4.2 (Functional impact of dyskinesias) in part IV from baseline to visit 4. Minimum score is 0 and maximum score is 8. A higher score means more dyskinesia.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mesdopetam | Placebo
Number analyzed (Participants) | 37 | 35
score on a scale | -1.3 [-1.8 to 0.8] | -0.6 [-1.1 to 0.1]

3. Secondary Outcome: Unified Parkinson's Disease Rating Scale (MDS-UPDRS), Part II and III
Description: Change in MDS-UPDRS sum score of parts II+III (Motor aspects of Experiences of Daily living + Motor Examination) from baseline to visit 4. Minimum value is 0 and maximum value is 124. Higher score mean a worse outcome.
Time Frame: Baseline and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Mesdopetam | Placebo
Number analyzed (Participants) | 37 | 35
score on a scale | -3.0 [-6.5 to 0.6] | -2.2 [-5.9 to 1.4]

4. Other Pre Specified Outcome: Change in Daily Hours Spent in ON-time With Troublesome Dyskinesia as Assessed by 24-hour Patient Diaries
Description: Change in ON-time with troublesome dyskinesia as assessed by patient completed 24-hour diaries, from run-in to visit 4. This is a self administered diary where patients assess their motor state every half hour during 24 hours.
  The different motor states assessed: ON, ON with troublesome dyskinesia, OFF and asleep.
Time Frame: Run-in and 4 weeks
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: daily hours
Arm/Group | Mesdopetam | Placebo
Number analyzed (Participants) | 37 | 34
daily hours | -3.3 [-4.3 to -2.4] | -1.7 [-2.8 to -0.7]

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Mesdopetam | Placebo
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/36
Other Adverse Events (participants affected / at risk) | 29/39 | 28/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mesdopetam (N=39) | Placebo (N=36)
Dizziness (Nervous system disorders) | 2 | 3
Dyskinesia (Nervous system disorders) | 4 | 2
Freezing phenomenon (Nervous system disorders) | 1 | 4
Headache (Nervous system disorders) | 5 | 5
On and off phenomenon (Nervous system disorders) | 2 | 1
Parkinsonism (Nervous system disorders) | 9 | 3 — In the mesdopetam group, 7 of the parkinsonism adverse events occurred during the titration phase (i.e. the first 2 weeks of study treatment) and only 2 of the parkinsonism event during steady state (i.e. the last 2 weeks of study treatment).
Fatigue (General disorders) | 2 | 9
Gait disturbance (Nervous system disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 2
Sleep disorder (Psychiatric disorders) | 3 | 2
Muscle spasm (Musculoskeletal and connective tissue disorders) | 0 | 2
Muscoloskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3
Nausea (Gastrointestinal disorders) | 0 | 4
Fall (Injury, poisoning and procedural complications) | 4 | 3
Urinary tract infection (Infections and infestations) | 2 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
There were technical difficulties in the administration of UDysRS objective score. It was not administered in a manner that would enable an unambiguous interpretation of the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-01-14): https://cdn.clinicaltrials.gov/large-docs/70/NCT03368170/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT03368170/SAP_001.pdf